CLINICAL TRIAL: NCT01965080
Title: Phase 2 Study of Exemestane in Advanced and Recurrent Endometrial Carcinoma
Brief Title: Exemestane in Advanced and Recurrent Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSGO-EC-0302
Record Dates: First submitted 2013-09-26; First posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exemestane (Experimental): Exemestane 25 mg daily
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Exemestane — One tablet Exemestane 25 mg daily
  Other Names: Aromasin

SUMMARY:
A phase II study of Exemestane in Advanced or recurrent endometrial carcinoma

Hypothesis: Treatment With Exemestane can give a response rate of at least 30%

DETAILED DESCRIPTION:
Patients With Advanced or recurrent endometrial cancer of endometrioid type were treated With Exemestane tablets 25 mg daily.

Patients were grouped according to estrogen receptor status.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent endometrial cancer not considered for treatment modalities apart from hormonal treatment
* Endometrioid histology
* Age above 18 years
* Post menopausal status
* Performance status 0-2
* Informed consent

Exclusion Criteria:

* Congestive heart disease grade III.IV
* History of thromboembolic signs
* Other primary hormonal therapy
* Patients With symptomatic brain metastasis
* Severe hepatic or renal impairment
* Pregnancy, lactation or child bearing potential without adequate contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months
  Objective response rate within 6 months of treatment

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Special attention to progression status at 6 months

OTHER OUTCOMES:
Toxicity | Up to 2 years
  Asses toxicity to the treatment using Common Toxicity Criteria for Adverse Effects

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Kristensen, MD, PhD, Study Chair — NSGO
Locations (1):
- The Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Derived] Lindemann K, Malander S, Christensen RD, Mirza MR, Kristensen GB, Aavall-Lundqvist E, Vergote I, Rosenberg P, Boman K, Nordstrom B. Examestane in advanced or recurrent endometrial carcinoma: a prospective phase II study by the Nordic Society of Gynecologic Oncology (NSGO). BMC Cancer. 2014 Feb 5;14:68. doi: 10.1186/1471-2407-14-68. PMID 24498853